CLINICAL TRIAL: NCT07139015
Title: Comparative Effects of Mirror Therapy and Constraint-induced Movement Therapy on Grip Strength, Hand Dexterity, and Upper Limb Motor Function in Post-stroke Patients.
Brief Title: Comparing Mirror Therapy and CIMT for Hand and Arm Function in Post-Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0283
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy; Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-Induced Movement Therapy (Experimental): Constraint-Induced Movement Therapy (CIMT) will involve placing a mitt or sling on the unaffected upper limb to promote use of the affected arm. Participants will attend sessions 5 days a week for 6 weeks, each lasting 60-90 minutes.
  Exercises include:
  Squeezing therapy putty (3 sets of 10-15 reps) Isometric grip holds (3 sets of 5-10 seconds) Finger-tapping (3 sets of 10 reps) Buttoning and zipping tasks (3 sets of 5-10 reps) The intervention targets grip strength, endurance, dexterity, and functional motor recovery through moderate-intensity, task-specific training.
  Interventions: Other: CONSTRAINT-INDUCED MOVEMENT THERAPY
- MIRROR THERAPY (Experimental): The experimental group will receive Mirror Therapy for 15-20 minutes per session, 5 days a week for 6 weeks. A mirror will be placed to reflect movements of the unaffected limb, creating the illusion that the affected limb is moving. Participants will perform simulated grasping, finger tapping, pegboard tasks, and wrist movements to engage mirror neurons and promote motor recovery.
  Interventions: Other: MIRROR THERAPY

INTERVENTIONS:
Other: CONSTRAINT-INDUCED MOVEMENT THERAPY — Constraint-Induced Movement Therapy (CIMT) involves restricting the unaffected arm to promote use of the affected limb through task-specific exercises. It is delivered 5 days a week for 6 weeks, with sessions lasting 60-90 minutes, focusing on improving strength, dexterity, and function.
  Arms: Constraint-Induced Movement Therapy
Other: MIRROR THERAPY — Mirror Therapy (MT) uses a mirror to reflect movements of the unaffected limb, creating the illusion of movement in the affected limb.
  Participants will do 60-90 minute sessions, 5 days a week for 6 weeks.
  Exercises include hand opening/closing, finger movements, and simple object tasks to improve motor function and coordination through visual feedback.
  Arms: MIRROR THERAPY

SUMMARY:
The goal of this clinical trial is to find out whether Mirror Therapy (MT) combined with Constraint-Induced Movement Therapy (CIMT) improves hand and arm function after a stroke. The study will also compare this combination to CIMT alone. The main questions it aims to answer are:

Does combining MT with CIMT improve grip strength, hand dexterity, and upper limb function more than CIMT alone? Which therapy is more effective in helping stroke survivors regain use of their arm and hand?

Participants will:

Be randomly assigned to receive either CIMT alone or CIMT combined with MT Attend therapy sessions 5 days a week for 6 weeks, each lasting 60-90 minutes Undergo tests before and after treatment to measure grip strength, dexterity, and motor function using tools like the Fugl-Meyer Assessment, Box and Block Test, and Hand-Held Dynamometer

DETAILED DESCRIPTION:
This randomized clinical trial aims to evaluate and compare the effects of Mirror Therapy (MT) and Constraint-Induced Movement Therapy (CIMT) on grip strength, hand dexterity, and upper limb motor function in post-stroke patients. Stroke is a leading cause of long-term disability, particularly affecting upper limb motor function, which severely impacts the ability to perform daily activities. This study seeks to provide insights into which approach or combination of therapies is more effective in improving upper limb functionality in post-stroke patients, thereby enhancing their quality of life and rehabilitation outcomes.

In this study, a randomized clinical trial (RCT) methodology will be utilized. 32 participants male and female patients aged 40 years and above who have a confirmed diagnosis of stroke, verified through CT scan and MRI imaging will be included. Eligible participants will have experienced a stroke within the past six months to ensure relevance to the intervention and recovery phase. Additionally, only those with a Brunnstrom grade of 2 or higher, indicating some degree of voluntary motor function, will be included by using non-probability convenience sampling and randomly divided into two groups: one receiving only CIMT and the other combining MT with CIMT. Baseline measurements will be taken for all participants to assess grip strength, hand dexterity, and upper limb motor function, utilizing validated tools like the Fugl-Meyer Assessment (FMA), Motor Activity Log (MAL), Box and Block Test (BBT), and Hand-Held Dynamometer. Both groups will undergo therapy sessions five days a week for six weeks, with daily sessions lasting 60-90 minutes. The data analysis will be performed using SPSS version 25. Data normality will be checked via the Shapiro-Wilk test. To evaluate within-group changes between pre- and post-treatment measurements, the Wilcoxon signed-rank test will be used, as it is appropriate for non-parametric data. The Mann-Whitney U test, a non-parametric test for comparing two independent groups.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Age 40 years and above
* Diagnosed patients confirmed by CT scan and MRI
* History of stroke not more than 6 months
* Brunnstrom grade 2 and above

Exclusion Criteria:

* Patients having history of musculoskeletal disorders
* History of shoulder injuries or adhesive capsulitis
* Patients having visual and auditory deficit will be excluded
* Patients who have sensory deficit will be excluded

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Grip strength | Baseline and after 6 weeks of intervention
  Change in grip strength of the affected hand, measured using a Hand-Held Dynamometer.
Hand dexterity | Baseline and after 6 weeks of intervention
  Change in fine motor skills assessed using the Box and Block Test (BBT).
Upper limb motor function | Baseline and after 6 weeks of intervention
  Improvement in overall motor function of the affected upper limb, assessed using the Fugl-Meyer Assessment (FMA) and Motor Activity Log (MAL).

CONTACTS AND LOCATIONS:
Overall Officials: HAMZA NAFEES, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Evercare Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No